CLINICAL TRIAL: NCT04272983
Title: Study of the Prevalence of Gluten-dependent Diseases in the Russian Population and the Development of New Biotechnological Approaches to Obtain Gluten-free Products
Brief Title: Population Study of the Prevalence of Celiac Disease and Other Gluten-dependent Disorders in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-15-10410
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-03

CONDITIONS: Celiac Disease in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To study the prevalence and clinical features of celiac disease in children to develop new treatment approaches and rehabilitation strategies.

DETAILED DESCRIPTION:
The purpose of this screening program is to identify people at high risk for developing celiac disease, which is due to the genetic intolerance of gluten - a protein found in wheat, rye and barley. When a person with celiac disease consumes gluten-containing foods, his immune system damages the mucous membrane of the small intestine. Inflammation develops and, as a result, the absorption of vitamins, minerals and other vital nutrients is disrupted. Studies have shown that timely diagnosis of celiac disease is important for the treatment or prevention of its complications. Left untreated, the disease can lead to impaired growth and development, diabetes, cancer, or other diseases. In Europe and the USA, celiac disease is a chronic disease that occurs in approximately one in 100 and one in 22 who have risk factors. There are frequent cases of an erased or low-symptom course of celiac disease. Unfortunately, ninety-seven percent of cases remain undiagnosed and, accordingly, do not receive proper treatment. A screening program will increase knowledge about the disease and contribute to the early detection of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Schoolchildren from various districts of Moscow selected as a result of questioning in the risk group for the development of celiac disease
* Availability of written informed consent of the child over 14 years of age to participate in the study;
* Availability of written informed consent of the parent of the child to participate in the study;
* Age from 7 to 18 years;
* Male and female gender;
* The number of points according to the results of the survey is more than 25.

Exclusion Criteria:

* Age up to 7 years and over 18 years.
* The lack of written informed consent of the child over 14 years of age to participate in the study;
* The lack of written informed consent of the parent / guardian of the child to participate in the study;
* The number of points on the results of the survey from 0 to 24

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Schoolchildren of the city of Moscow
Sampling Method: Non-Probability Sample
Enrollment: 3070 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Questioning of schoolchildren | 2 year
  Questionnaire by specially developed questionnaire. A structured questionnaire was used to collect data on symptoms and signs that are known to be associated with celiac disease. Each of the following statements begin with "Does your child have ...? " Scoring: Never=1; Seldom= 2; Frequent=3; A Lot=4; Don't Know=0; No=1; Yes=2 If the total score was 25 or more, then this respondent belongs to the high risk group for the development of celiac disease.
Serological and genetic studies at risk group | 3 year
  Serological and genetic testing in the laboratory. Screening for celiac disease for suspected celiac disease carried out by testing in an independent laboratory serological examinations (total IgA, AT to tissue transglutaminase IgA, AT to tissue transglutaminase IgG, AT to endomysium IgA); genetic screening - HLA-DQ2 / DQ8; IgE (wheat flour, F4).

CONTACTS AND LOCATIONS:
Overall Officials: Svetlana Erdes, Ph.D, Study Chair — Sechenov First Moscow State Medical University
Locations (1):
- Erdes Svetlana, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
The local ethics committee does not allow. But upon official request can provide.

REFERENCES:
- [Background] Savvateeva LV, Erdes SI, Antishin AS, Zamyatnin AA Jr. Overview of Celiac Disease in Russia: Regional Data and Estimated Prevalence. J Immunol Res. 2017;2017:2314813. doi: 10.1155/2017/2314813. Epub 2017 Feb 20. PMID 28316996
- [Background] Savvateeva LV, Erdes SI, Antishin AS, Zamyatnin AA Jr. Current Paediatric Coeliac Disease Screening Strategies and Relevance of Questionnaire Survey. Int Arch Allergy Immunol. 2018;177(4):370-380. doi: 10.1159/000491496. Epub 2018 Jul 27. PMID 30056445
- [Background] Lototskaya PS, Manina MA, Tertychnyy AS, Zamyatnin AA Jr, Erdes SI. Duodenal Ulceration in a Child with Coeliac Disease. Diagnostics (Basel). 2020 Jan 9;10(1):31. doi: 10.3390/diagnostics10010031. PMID 31936445